CLINICAL TRIAL: NCT05057312
Title: Promoting HPV Vaccination Among Young Adults in Texas
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Prevention
Other Study IDs: 2020-1142; R01CA248216 (NIH); NCI-2021-09416 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-1142 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2021-08-25; First posted 2021-09-27 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Human Papillomavirus Infection
MeSH Terms: conditions — Papillomavirus Infections | interventions — Interviews as Topic

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Group I (standard CDC information) (Active Comparator): Participants receive standard CDC information about HPV vaccination.
  Interventions: Other: Informational Intervention; Other: Interview; Other: Questionnaire Administration
- Group II (video narratives) (Experimental): Participants receive video narratives about HPV vaccination.
  Interventions: Other: Informational Intervention; Other: Interview; Other: Questionnaire Administration
- Group III (written narratives) (Experimental): Participants receive written narratives about HPV vaccination.
  Interventions: Other: Informational Intervention; Other: Interview; Other: Questionnaire Administration
- Group IV (enhanced access to vaccine, CDC information) (Experimental): Participants receive enhanced access to vaccination and standard CDC information about HPV vaccination.
  Interventions: Other: Enhancing Accessibility to Health Care; Other: Informational Intervention; Other: Interview; Other: Questionnaire Administration
- Group V (enhanced access to vaccine, video narratives) (Experimental): Participants receive enhanced access to vaccination and video narratives about HPV vaccination.
  Interventions: Other: Enhancing Accessibility to Health Care; Other: Informational Intervention; Other: Interview; Other: Questionnaire Administration
- Group VI (enhanced access to vaccine, written narratives) (Experimental): Participants receive enhanced access to vaccination and written narratives about HPV vaccination.
  Interventions: Other: Enhancing Accessibility to Health Care; Other: Informational Intervention; Other: Interview; Other: Questionnaire Administration

INTERVENTIONS:
Other: Enhancing Accessibility to Health Care — Receive enhanced access to vaccination
  Arms: Group IV (enhanced access to vaccine, CDC information); Group V (enhanced access to vaccine, video narratives); Group VI (enhanced access to vaccine, written narratives)
Other: Informational Intervention — Receive standard CDC information
  Arms: Group I (standard CDC information); Group IV (enhanced access to vaccine, CDC information)
Other: Informational Intervention — Receive video narratives
  Arms: Group II (video narratives); Group V (enhanced access to vaccine, video narratives)
Other: Informational Intervention — Receive written narratives
  Arms: Group III (written narratives); Group VI (enhanced access to vaccine, written narratives)
Other: Interview — Ancillary studies
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
This clinical trial studies how to improve the human papillomavirus (HPV) vaccination rate in young adults in Texas. This trial aims to learn more about how researchers and health care providers can increase HPV vaccination among college students.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the impact of addressing individual and system levels of influence on HPV vaccination initiation and completion rates.

II. To gain insight into mechanisms of the intervention's efficacy, individual differences, and implementation of the intervention using mixed methods.

OUTLINE: Participants are randomized to 1 of 6 groups.

GROUP I: Participants receive standard Centers for Disease Control and Prevention (CDC) information about HPV vaccination.

GROUP II: Participants receive video narratives about HPV vaccination.

GROUP III: Participants receive written narratives about HPV vaccination.

GROUP IV: Participants receive enhanced access to vaccination and standard CDC information about HPV vaccination.

GROUP V: Participants receive enhanced access to vaccination and video narratives about HPV vaccination.

GROUP VI: Participants receive enhanced access to vaccination and written narratives about HPV vaccination.

After completion of study, participants are followed up at 3 and 9 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-26 years. This criterion is based on the CDC recommendation of vaccination up to 26 years of age and the fact that individuals 18 years and older can consent by themselves for on-site vaccination
* Ability to read and understand English
* Self-identification as not yet having received any HPV vaccine injections. Self-identification is justified because it is safe to be vaccinated again, which could happen if a previously vaccinated person forgets their vaccination. Furthermore, in a person previously vaccinated with an older version of the vaccine, which targeted fewer HPV types, receiving the newer version would be advantageous and not cause any harm. Alternatives to self-identification, such as obtaining medical records from doctors' offices, would be very challenging for young adults, especially for those who do not remember when and where they might have received vaccination
* Access to a smart phone, tablet or computer that is connected to the internet
* Current enrollment in one of the participating schools with an anticipated continuous enrollment of at least 9 months

Exclusion Criteria:

* Being pregnant
* Having a life-threatening allergy to any component of the HPV vaccine

Ages: 18 Years to 26 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1200 (Estimated)
Dates: Start 2021-07-26 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Rate of human papillomavirus (HPV) vaccination initiation | At 3 months
Rate of HPV vaccination completion | At 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Qian Lu, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Lu Q, Dawkins-Moultin L, Cho D, Tan NQP, Hopfer S, Li Y, Ramondetta L, Xu Y, Lun D, Chen M. A multilevel intervention to promote HPV vaccination among young adults in Texas: protocol for a randomized controlled trial. BMC Public Health. 2024 Jun 5;24(1):1506. doi: 10.1186/s12889-024-18828-9. PMID 38840086